CLINICAL TRIAL: NCT02394756
Title: Investigation of Ocular Signs & Symptoms in Wearers Fitted With Contact Lenses Following Digital Device Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-5615
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2017-03

CONDITIONS: Visual Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Marketed Soft Contact Lens (Test) (Experimental): Subjects will be randomized to wear each of three contact lens types (Marketed Soft Contact lens, AIR OPTIX® AQUA, or Biofinity®) for a 4-week period with each lens type.
  Interventions: Device: Marketed Soft Contact lens; Device: AIR OPTIX® AQUA; Device: Biofinity®
- AIR OPTIX® AQUA (Active Comparator): Subjects will be randomized to wear each of three contact lens types (Marketed Soft Contact lens, AIR OPTIX® AQUA, or Biofinity®) for a 4-week period with each lens type.
  Interventions: Device: Marketed Soft Contact lens; Device: AIR OPTIX® AQUA; Device: Biofinity®
- Biofinity® (Active Comparator): Subjects will be randomized to wear each of three contact lens types (Marketed Soft Contact lens, AIR OPTIX® AQUA, or Biofinity®) for a 4-week period with each lens type.
  Interventions: Device: Marketed Soft Contact lens; Device: AIR OPTIX® AQUA; Device: Biofinity®

INTERVENTIONS:
Device: Marketed Soft Contact lens — Replacement schedule every 2 weeks
  Other Names: senofilcon A
Device: AIR OPTIX® AQUA — Replacement schedule every 4 weeks
  Other Names: lotrafilcon B
Device: Biofinity® — Replacement schedule every 4 weeks
  Other Names: comfilcon A

SUMMARY:
The objective of this study is to assess how various silicone hydrogel lenses perform when worn by subjects who are heavy digital device users.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand and sign the statement of Informed Consent and receive a fully executed copy of the form.
2. The subject must be between 18 and 40 years of age.
3. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -0.50D to -8.00D in each eye.
4. The subject's refractive cylinder must be no more than -1.25 D cylindrical correction in each eye after vertexing to the corneal plane.
5. The subject must have best corrected visual acuity of 0.20 or better in each eye.
6. The subject must be a current wearer of daily, spherical, soft contact lenses (no bifocal or multifocal contact lenses, no extended wear or monovision) for at least 5 days/ week and at least 8 hours/day during the month prior to enrollment.
7. The subject must be using digital devices (any combination of computers, tablets, smartphones, etc.) for at least 8 hours over the course of a typical day.
8. The subject should own a wearable pair of spectacles and wear them the day of the baseline visit.
9. The subject must have normal eyes with no evidence of abnormality or disease that in the opinion of the investigator would contraindicate contact lens wear.
10. The subject must meet normal eligibility conditions of binocular vision tests.
11. The subject may not have any double vision at near with their habitual contact lens correction.

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear (at the investigator's discretion).
3. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear (at the investigator's discretion).
4. Use of any medication that causes side effects similar to side effects experienced when using digital devices, such as subjects reporting headaches associated with birth control pills (at the investigator's discretion).
5. Any infectious disease (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease.
6. Any active ocular infection.
7. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by keratometry.
8. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.).
9. Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
10. Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
11. Any known hypersensitivity or allergic reaction to the study products.
12. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
13. History of binocular abnormality or strabismus.
14. Employee of investigational clinic (e.g. Investigator, Coordinator, Technician).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 52 subjects were enrolled in this study. Of the enrolled subjects 10 subjects did not meet the eligibility criteria and 42 subjects were dispensed study lenses. Of the dispensed subjects 37 completed the study while 5 subjects were discontinued.
Groups:
- Senofilcon A/Lotrafilcon B/Comfilcon A: Subjects randomized to this sequence wore the senofilcon A lens in the first period, the lotrafilcon B lens in the second period and the comfilcon A lens in the third period.
- Senfilcon A/Comfilcon A/Lotrafilcon B: Subjects randomized to this sequence wore the senofilcon A lens in the first period, the comfilcon A lens in the second period and the lotrafilcon B lens in the third period.
- Lotrafilcon B/Comfilcon A/Senofilcon A: Subjects randomized to this sequence wore the lotrafilcon B lens in the first period, the comfilcon A lens in the second period and the senofilcon A lens in the third period.
- Lotrafilcon B/Senofilcon A/Comfilcon A: Subjects randomized to this sequence wore the lotrafilcon B lens in the first period, the senofilcon A lens in the second period and the comfilcon A lens in the third period.
- Comfilcon A/Senofilcon A/ Lotrafilcon B: Subjects randomized to this sequence wore the comfilcon A lens in the first period, the senofilcon A lens in the second period and the lotrafilcon B lens in the third period.
- Comfilcon A/Lotrafilcon B/Senofilcon A: Subjects randomized to this sequence wore the comfilcon A lens in the first period, the lotrafilcon B lens in the second period and the senofilcon A lens in the third period.
Period: Period 1
Arm/Group | Senofilcon A/Lotrafilcon B/Comfilcon A | Senfilcon A/Comfilcon A/Lotrafilcon B | Lotrafilcon B/Comfilcon A/Senofilcon A | Lotrafilcon B/Senofilcon A/Comfilcon A | Comfilcon A/Senofilcon A/ Lotrafilcon B | Comfilcon A/Lotrafilcon B/Senofilcon A
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 6 | 6 | 6 | 7 | 6
Not Completed | 0 | 1 | 1 | 1 | 0 | 1
Not completed — Lens Discomfort | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 0 | 0
Period: Period 2
Arm/Group | Senofilcon A/Lotrafilcon B/Comfilcon A | Senfilcon A/Comfilcon A/Lotrafilcon B | Lotrafilcon B/Comfilcon A/Senofilcon A | Lotrafilcon B/Senofilcon A/Comfilcon A | Comfilcon A/Senofilcon A/ Lotrafilcon B | Comfilcon A/Lotrafilcon B/Senofilcon A
Started | 7 | 6 | 6 | 6 | 7 | 6
Completed | 7 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Unsatisfactory Visual Response | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 3
Arm/Group | Senofilcon A/Lotrafilcon B/Comfilcon A | Senfilcon A/Comfilcon A/Lotrafilcon B | Lotrafilcon B/Comfilcon A/Senofilcon A | Lotrafilcon B/Senofilcon A/Comfilcon A | Comfilcon A/Senofilcon A/ Lotrafilcon B | Comfilcon A/Lotrafilcon B/Senofilcon A
Started | 7 | 6 | 6 | 6 | 6 | 6
Completed | 7 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least one study lens.
Groups:
- Dispensed Subjects: All subjects that were dispensed at least 1 study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (4.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 20
  Black or African American | 1
  White | 21
Region of Enrollment [Number; unit: participants]
  Canada | 42

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Comfort
Description: Subjective Overall Comfort was evaluated using the Contact Lens User Experience Comfort scores (CLUE). CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. Scores range 0-120.
Time Frame: 1-Day Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Senofilcon A: Subjects wore the senofilcon A lens in any of the three periods during the study.
- Lotrafilcon B: Subjects wore the lotrafilcon B lens in any of the three periods during the study.
- Comfilcon A: Subjects wore the comfilcon A lens in any of the three periods during the study.
Arm/Group | Senofilcon A | Lotrafilcon B | Comfilcon A
Number analyzed (Participants) | 37 | 37 | 37
units on a scale | 65.0 (19.76) | 53.6 (23.34) | 61.9 (22.70)

2. Primary Outcome: Subjective Overall Quality of Vision
Description: Subjective Overall quality of vision was evaluated using the Contact Lens User Experience Comfort scores (CLUE). CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. Scores range 0-120.
Time Frame: 1-Day Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Senofilcon A | Lotrafilcon B | Comfilcon A
Number analyzed (Participants) | 37 | 37 | 37
units on a scale | 63.6 (17.76) | 63.8 (18.24) | 65.8 (18.39)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 4-weeks per subject.
Arm/Group | Senofilcon A | Lotrafilcon B | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 3/42 | 0/42 | 2/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon A (N=42) | Lotrafilcon B (N=42) | Comfilcon A (N=42)
Non-Significant Infiltrate Event (Eye disorders) | 3 (5) | 0 (0) | 2 (2)
Common Cold (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) — Not study related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days